# A Single Center, Randomized, Double-Blind Controlled Trial of Sitagliptin Versus Placebo to Reduce the Incidence and Severity of New-onset Diabetes After Kidney Transplant

## March 11, 2015 Protocol # 50669 Version 6

## Study protocol and Statistical Analysis Plan

## Inclusion/Exclusion

#### Inclusion criteria

- 1. Adult (≥18 yo) recipient of living-donor or deceased donor kidney transplant
- 2. Blood sugar ≥ 200 mg/dL in first 120 hours after transplant
- 3. No history of diabetes or prior treatment with insulin or oral hypoglycemic agents

#### Exclusion criteria

- 1. A1c of ≥6.5% measured immediately pre-transplant
- 2. Recipient of simultaneous kidney-pancreas, kidney-liver, kidney-heart, or kidney-lung transplant
- 3. Prior non-renal solid organ transplant

## Study procedures

## Sitagliptin dosing

In patients randomized to sitagliptin, the initial dose will be 100mg oral per day, adjusted based on creatinine clearance per prescribing information (9):

| Creatinine clearance (mL/min) | Sitagliptin dose (mg orally per day) |
|-------------------------------|--------------------------------------|
| ≥ 50 | 100 |
| ≥30 and <50 | 50 |
| <30 or on dialysis | 25 |

Screening period (Visit 1)

All patients presenting for living-donor or deceased donor kidney transplant will have a medical history, medication history, vital signs, height, weight, body mass index, physical exam, random blood sugar, HbA1c and EKG done as part of routine pre-transplant protocol at Barnes Jewish Hospital. Patients with hyperglycemia, defined as a random blood sugar ≥ 200 mg/dL, in the first 120 hours after kidney transplant will be screened to determine eligibility for the study based on inclusion and exclusion criteria.

#### Randomization (Visit 2)

Patients meeting study entry criteria and consenting to study participation will be stratified based on HbA1c (<5.7 or 5.7-6.4%) and block randomized in blocks of eight in a 1:1 ratio to sitagliptin versus placebo. Sitagliptin dose will be 100mg/day, adjusted per creatinine clearance and tolerability. A fasting blood sugar will be obtained prior to initiation of sitagliptin. Patients will be instructed by a licensed diabetic educator on proper measurement and recording of fasting and post-prandial blood sugars. Subjects will be provided a log, standard glucometer and testing strips to maintain a blood sugar log post-discharge. Visit 2 will occur within 24 hours after Visit 1.

## Drug dosing period (Visits 3-4)

Sitagliptin or placebo will be continued until 3 months post-transplant, at which time study medication will be discontinued and collected from the subject. At the 1 and 3 month visits, vital signs, height, weight, and BMI will be obtained. A physical exam will be performed. Blood sugar logs provided by the patient will be reviewed and adverse effects recorded. At the 3 month visit (Visit 4), a HbA1c, 2-hour OGTT, fasting C-peptide and insulin level will be obtained.

#### Follow-up (Visit 5)

At the 6 month final visit, 3 months following discontinuation of study medication, vital signs, height, weight, BMI, HbA1c, 2-hour OGTT, fasting C-peptide and insulin level will be obtained. A physical exam will be performed. Blood sugar logs provided by the patient will be reviewed and adverse effects recorded.

## **Efficacy Assessment**

## Efficacy assessment

Efficacy of sitagliptin versus placebo in 1) lowering 2-hour OGTT by  $\geq$  20 mg/dL, 2) preventing NODAT defined by normal 2-hour OGTT and 3) improving HbA1c by  $\geq$ 0.5% will be assessed at 3 months post-transplant.

## Statistical analysis

The following testing methods will be used in the study:

# Statistical methods

Oral Glucose tolerance test - T-test or Mann-Whitney U

Hemoglobin A1c - T-test or Mann-Whitney U

# Power/Sample size:

Based on a sample size of 25 patients per group, this study has over 80.7% power to detect a difference of 20 mg/dL in 2-hour OGTT. This calculation assumes a standard deviation of 25 mg/dL or less between groups. However to account for study drop out and loss to follow-up (those who did not take study drug or did not come for follow-up), the study expanded to include 61 patients.